CLINICAL TRIAL: NCT02249312
Title: The Effect of BIIL 284 BS (14 Day Treatment) on Induced-sputum Variables in Patients With Bronchial Asthma (a Double-blind, Randomized, Placebo-controlled Parallel Study)
Brief Title: The Effect of BIIL 284 BS on Induced-sputum Variables in Patients With Bronchial Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.11
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — amelubant

ARMS (2):
- BIIIL (Experimental)
  Interventions: Drug: BIIL 284 BS
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS
  Arms: BIIIL
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate the anti-inflammatory effect of BIIL 284 BS compared with placebo in patients with asthma

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated prior to participation into the study
* Males and females aged 18 - 65 years. Female patients of child bearing potential cannot participate in this study. Female patients are eligible to participate only if they are surgically sterilized or two years post menopausal. Women entering into this trial will have a pregnancy test before and after participation in the trial. Testing will be done during visit 1 and visit 5
* A documented diagnosis of asthma as defined by the American thoracic society i.e., episodic wheezing, chest tightness, cough and/or shortness of breath at least partially relieved by bronchodilator medication. No hospital admission in the last eight weeks for the treatment of asthma; no requirement for steroid therapy (systemic or inhaled) for the previous four weeks, nedocromil sodium or sodium cromoglycate in the previous two weeks; asthma therapy stable and limited to intermittent use of inhaled β2-agonists or anticholinergics on an as required basis, or occasional use of antihistamines. Predicted equations for forced expiratory volume in one second (FEV1) of Caucasians and African - Americans are those of Morris et. al. and Glindmeyer et. al. At visit 2, 3, and 5, immediately prior to the induced sputum test, but following albuterol administration, a patient's FEV1 must be above 60 % of predicted
* The presence of, at least, 25 % of neutrophils in induced sputum during screening visit 2 (this requirement refers to the neutrophils percentage exclusive of squamous cells)
* Ability to produce an adequate induced sputum sample (visit 2) as defined by: Volume > 1 ml, squamous cells < 80 % and ability to tolerate the procedure for at least 4 minutes with no bronchoconstriction (a fall in FEV1 > 20 %)
* Patients with PC20 methacholine <= 8 mg/ml as determined at visit 1
* Non-smokers (patients who have never smoked) or ex-smokers for at least one year with a smoking history, no greater than five pack-years (1 pack year = 20 cigarettes per day for 1 year)
* Ability to be trained in the proper use of peak flow meter (Mini Wright peak flow meter, Clement Clarke, Inc.) and in performing and recording technically satisfactory pulmonary function tests
* Willing to attend an outpatient clinic on a regular basis and undergo three induced sputum challenges during which they will be confined to the investigational unit for up to two hours
* Ability to comply with the concomitant therapy restrictions
* Patients will be off all prescription drug therapy other than that specifically for asthma or hay fever. Over the counter (O.T.C.) drugs must be discontinued for at least two weeks prior to participation in the study. If any O.T.C. medication is needed by patients throughout the study, the investigator will call the clinical monitor and this will be reviewed on a case-by-case basis
* Patients will have no evidence of clinically relevant concomitant disease based upon complete medical history, full physical examination, chest x-ray (if not done in previous 6 months), electrocardiogram (ECG) and clinical laboratory tests. These tests should indicate that the patient is healthy except for changes related to asthma or atopy (e.g., eosinophilia based on a total eosinophil count). Patient may have a history of allergic rhinitis or urticaria.

  * The following laboratory parameters must be within the normal range, or if not, be documented by the investigator as not clinically relevant:
  * Routine urinalysis, Complete blood cell (CBC) (excluding White blood cell (WBC)) , Na, K, Ca, Cl, Gamma-glutamyl-transferase (GGT), Lactic dehydrogenase (LDH), bicarbonate, inorganic phosphorus, glucose, uric acid, triglyceride, total protein, albumin and cholesterol.
  * The following test may be outside the normal range to the extent indication:

    * Test a; Liver function tests: serum glutamic oxaloacetic transaminase / aspartate aminotransferase (SGOT/AST), serum glutamic pyruvic transaminase / alanine transaminase (SGPT/ALT), total bilirubin (in patients with an isolated raised bilirubin and diagnosis of " suspected Gilbert's syndrome" will be accepted only after the effect of high carbohydrate meal or bilirubin level has been determined) and alkaline phosphatase with a cut off for exclusion by 10 % > ULN (upper limit of normal range for the measuring laboratory)
    * Test b; Hematology: WBC with a cut off for exclusion by < 3.80 x 10**9 /L, neutrophils with a cut off for exclusion by < 2.00 x 10**9 /L, platelets with a cut off for exclusion by < 100 x 10**9 /L, hemoglobin with a cut off for exclusion by < 12 g/dL
    * Test c; urea nitrogen and creatinine with a cut off for exclusion by 10 % > ULN

Exclusion criteria:

* Viral respiratory tract infection, respiratory tract infection or asthma exacerbation within the six weeks preceding the study or, if hospitalized for their asthma in the last eight weeks
* Evidence of relevant concomitant disease based on complete medical history, full physical examination and clinical laboratory tests
* Known drug or alcohol dependence (absence of dependency for 10 years), history of significant allergic reactions to drugs or sensitivity to aspirin
* Use of an investigational new drug in the preceding month or six half lives (whichever is greater) prior to the first screen at visit 1
* Donate of blood during the preceding month of visit 1
* Patients receiving hyposensitization therapy who are not on a stable dose for the last three months before visit 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1999-07; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Percentage of neutrophils in induced sputum differential cell count | Baseline, Day 1 and 14

SECONDARY OUTCOMES:
Concentration of myeloperoxidase (MPO) in induced sputum | Baseline, Day 1 and 14
Concentration of Interleukin-8 (IL-8) in induced sputum | Baseline, Day 1 and 14
Concentration of tumor necrosis factor (TNF) alpha in induced sputum | Baseline, Day 1 and 14
Differential cell count in induced sputum | Baseline, Day 1 and 14
  eosinophils, basophils, macrophages, lymphocytes and epithelia cells
Changes in expression of Epidermal growth Factor (EGF) receptors in induced sputum | Day 1 and 14
  only in US center
Changes in expression of tissue growth factor (TGF) alpha in induced sputum | Day 1 and 14
  only in US center
Changes in expression of MUC5AC (maximum use concentration) in induced sputum | Day 1 and 14
  only in US center
Changes in forced expiratory volume in one second (FEV1) | Up to Day 27 after drug administration
  assessed by spirometry
Changes in forced vital capacity (FVC) | Up to Day 27 after drug administration
  assessed by spirometry
Changes in forced expiratory flow (FEF) 25-70% | Up to Day 27 after drug administration
  assessed by spirometry
Changes in FEF50% | Up to Day 27 after drug administration
  assessed by spirometry
Changes in FEF 75% | Up to Day 27 after drug administration
  assessed by spirometry
Changes in peak expiratory flow rate (PEFR) a.m. versus p.m.by patients daily records | Up to Day 27 after drug administration
Physician's global evaluation of symptoms assessed on a 6 point severity scale | Baseline, Day 14
Inhibition of MAC-1 expression | Day 1 and 14
Number of patients with Adverse Events | Up to day 27 after drug administration